CLINICAL TRIAL: NCT05187481
Title: Efficacy Evaluation of Jianpi Huatan Decoction in the Treatment of Advanced Colorectal Cancer and Analysis of Dominant Population Characteristics and Methylation Characteristics
Brief Title: Effect of Jianpi Huatan Decoction on Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: China Academy of Chinese Medical Sciences (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CI2021A01803
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-11

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal cancer; traditional Chinese medicine
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will take Jianpi Huatan dispensing granule while receiving chemotherapy and/or targeted therapy, once a day in the morning and evening, 30 days as a course of treatment, a total of 3 courses.
  Interventions: Drug: Jianpi Huatan dispensing granule
- Control Group (Placebo Comparator): The experimental group will take Placebo granule (containing 1/10 of the formula dose of Jianpi Huatan Granule) while receiving chemotherapy and/or targeted therapy, once a day in the morning and evening, 30 days as a course of treatment, a total of 3 courses.
  Interventions: Drug: Placebo granule

INTERVENTIONS:
Drug: Jianpi Huatan dispensing granule — once a day in the morning and evening, 30 days as a course of treatment, a total of 3 courses.
  Arms: Experimental Group
Drug: Placebo granule — once a day in the morning and evening, 30 days as a course of treatment, a total of 3 courses.
  Arms: Control Group

SUMMARY:
This study will take progression-free survival and overall survival as the main evaluation indexes, to evaluate the Efficacy of Jianpi Huatan Decoction in the Treatment of Advanced Colorectal Cancer. Decision Trees and Discriminant Analysis will be used to analyze the characteristics of dominant population combined with clinical data of patients. DNA methylation of the subjects will be detected to study the methylation characteristics of the preponderant population of Jianpi Huatan Decoction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with colorectal cancer with clear pathological diagnosis and Western medicine diagnostic criteria.
2. TNM classification of stage IV disease according to National Comprehensive Cancer Network (NCCN) Guidelines.
3. Expected survival time is over 3 months.
4. The age of 18 years old or more.
5. According to the efficacy evaluation criteria for solid tumors (RECIST 1.1), there are measurable lesions.
6. Chemotherapy and/or targeted therapy are planned.
7. Signed informed consent.

Exclusion Criteria:

1. History of previous or combined malignancies except non-melanoma skin cancer, cervical cancer in situ, or bladder cancer (Tis and T1) received adequate treatment in the five years prior to screening.
2. Combined with severe heart, liver, lung and kidney disease.
3. Patients have intestinal obstruction can't take decoction and need intravenous high-energy nutrition. Patients have malabsorption syndrome or other disease affecting gastrointestinal absorption or have active peptic ulcer disease.
4. Any unstable condition or condition that may endanger patient safety and compliance with research, such as pregnancy, depression, manic-depressive disorder, obsessive-compulsive disorder, or schizophrenia.
5. The expected survival time is less than 3 months.
6. The researchers determine that they were not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of randomization until the date of disease progression or date of death from any cause, whichever came first, assessed up to 100 months
  From enrollment until disease progression or death
Overall survival | From date of randomization until the date of death from any cause, assessed up to 100 months
  From enrollment until death or end of the follow-up

SECONDARY OUTCOMES:
Survival rate | 3 years
  The 1-year, 2-year and 3-year survival rates of patients in the treatment group and the control group were analyzed
Disease control rate | 3 months
  Efficacy was assessed according to RECIST 1.1 at the end of 3 months of treatment.
Cancer fatigue score | 3 months
  Piper Fatigue Scale will be used.The fatigue of patients will be evaluated from 22 items of behavioral dimension, emotional dimension, sensory dimension and cognitive dimension. The higher the score of each dimension, the more serious the fatigue degree.
Traditional Chinese Medicine(TCM )symptom grading table | 3 months
  Effective: after treatment, TCM symptom score decreased by more than 50% compared with that before treatment.
  Effective: decrease < 50% and equal to 30%; Invalid: decrease < 30%. Note: the formula is: (before treatment - integral after treatment) / before treatment by 100%.
The European Organization for Cancer Research and Treatment Core Quality of Life Questionnaire (EORTC QLQ-C30) score scale | 3 months
  The raw scores for the scales and single items were linearly transformed to values between 0 and 100 as described in the EORTC QLQ scoring manual. The mean and standard deviation of each scale/single item were calculated. A higher score for a functioning scale represented a healthier level of functioning, a higher score for the global health status scale represented a higher QOL, and a higher score for a symptom scale/item represented a worse level of symptomatology.
the United States Eastern Oncology Collaboration Group (ECOG) score scale | 3 months
  ECOG scoring standard is an indicator of patients' general health status and tolerance to treatment based on their physical strength. ECOG physical condition rating standard score 0-5 points. A minimum score of 0 indicates normal activity, a higher score indicates less physical activity, and a score of 5 indicates death.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Wu, Master, Study Chair — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided